CLINICAL TRIAL: NCT06742489
Title: Research for the Efficacy and Safety of Percutaneous Tibial Nerve Stimulation to Promote Storage Symptoms Postoperative Recovery for Patients With Benign Prostatic Hyperplasia(Randomised, Double-blind, Prospective, Single-centre Clinical Trial)
Brief Title: Research for the Efficacy and Safety of Percutaneous Tibial Nerve Stimulation to Promote Storage Symptoms Postoperative Recovery for Patients With Benign Prostatic Hyperplasia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhu Yiping (Other)
Responsible Party: Sponsor-Investigator, Zhu Yiping, Doctor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024218
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: This trial will include patients with storage symptoms as the main manifestation and undergo surgical treatment for benign prostatic hyperplasia. There is still a lack of similar products on the market to be used as a control, and thus the sham group will use the same device without therapeutic effect as a blank control.
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Participants in this group will receive T-PTNS three times a week for 30 minutes every time.
  Interventions: Device: Percutaneous tibial nerve stimulation device
- Sham group (Sham Comparator): The sham group will use the same device without therapeutic effect as a blank control.
  Interventions: Device: Sham group device

INTERVENTIONS:
Device: Percutaneous tibial nerve stimulation device — T-PTNS primarily delivers electrical stimulation to the sacral voiding center via the tibial nerve through the S2-S4 sacral plexus via skin-surface electrodes to improve patients' symptoms of urinary frequency, urgency, and urge incontinence.
  Arms: Treatment group
Device: Sham group device — The device in the sham group is manufactured by the same company and has the same appearance, display interface, and operation method as the device in the treatment group. These devices have the output circuit disconnected and no actual current output.
  Arms: Sham group

SUMMARY:
The goal of this clinical trial is to guide and promote the clinical application of T-PTNS in promoting the postoperative recovery of urinary storage symptoms in patients with BPH. The main question is to evaluate the effectiveness and safety of T-PTNS in promoting the improvement of postoperative urinary storage symptoms in patients with BPH through a single-center randomized double-blind controlled trial, and to propose standard parameters for use such as frequency and power, and ultimately to establish a standard process of T-PTNS treatment and form a replicable and promotable therapeutic specification. Participants will receive T-PTNS three times a week for 30 minutes every time. T-PTNS will be discontinued after 6 weeks. The study will last for 12 weeks, and subjects will be followed up periodically during the study period by the relevant researchers.

ELIGIBILITY:
Inclusion Criteria:

1. Participants have been fully informed of the potential benefits and risks associated with the trial and have provided written consent to participate.
2. Male participants between the ages of 45 and 80 are eligible to participate in the trial.
3. Participants with a confirmed diagnosis of Benign Prostatic Hyperplasia, a maximum urinary flow rate of ≤ 15 ml/sec, undergoing surgical treatment (Thulium laser vapoenucleation) and fulfilling any one of the following conditions according to the International Prostate Symptom Score (IPSS): a) any single IPSS urinary storage subscore (urinary frequency, urgency, nocturia frequency) greater than or equal to 3 points; b) a total IPSS storage subscore of 9 points or greater;
4. Participants who are able to discontinue relevant medications (M-blockers and β3 agonists) for a period of at least one week prior to enrolment;
5. Participants with autonomy, self-care, self-control, and the ability to use the toilet independently.

Exclusion Criteria:

1. Subjects presenting with urinary incontinence due to reduced sphincter function, or subjects evaluated for neurogenic bladder;
2. Subjects with urethral strictures or bladder neck contractures that make insertion of devices difficult;
3. Subjects with pacemakers, buried cardioverter-defibrillators, or other therapeutic electronic medical devices (including sacral neuromodulation).
4. Subjects with implanted devices in the body;
5. Subjects with untreated urinary tract infections;
6. Subjects with urinary stones that cause lower urinary tract symptoms;
7. Subjects with previous pelvic surgery; and
8. Subjects with a history of previous pelvic surgery, or colorectal surgery (except polypectomy and haemorrhoidectomy);
9. Subjects with untreated malignant tumors;
10. Subjects with neurological or cerebrovascular lesions or injuries, or medical conditions affecting cognition, bladder function, sphincter function, or urethral muscle function;
11. Subjects with skin breakdown, malignant tumors, or acute purulent inflammation on the surface of the plantar foot at the location where the electrode pads are to be placed;11. Subjects who have participated in a clinical trial of another drug within three months or a clinical trial of another medical device within 30 days;
12. Other conditions that the investigator deems unsuitable for participation in the study.

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptoms Score improvement percentage | 2,4,6,8,12 weeks after surgery
  The study will use International Prostate Symptoms Score (IPSS) questionnaire to evaluate the effectiveness of the treatment. IPSS improvement percentage is defined as dividing the difference between preoperative and postoperative IPSS by preoperative IPSS, which varies from 0% to 100%. If the score is over 50%, the treatment will be considered as effective.
Quality of Life change | 2,4,6,8,12 weeks after surgery
  The study will use International Prostate Symptoms Score (IPSS) questionnaire to evaluate the effectiveness of the treatment. Quality of Life (QoL) is the last question of the questionnaire. QoL change is defined as the difference between preoperative and postoperative QoL, which varies from 0 to 6. If the score is over 3, the treatment will be considered as effective.

SECONDARY OUTCOMES:
maximum urinary flow change | 6,12 weeks after surgery
  The study will use free uroflow to assess objective change, with maximum urinary flow (Qmax) as the primary outcome measure. Qmax change is defined as the difference between preoperative and postoperative Qmax. The score is not capped, but the higher the score, the better the outcome.
Overactive Bladder Symptom Score change percentage | 2,4,6,8,12 weeks after surgery
  The study will use Overactive Bladder Symptom Score (OABSS) questionnaire to evaluate the effectiveness of the treatment. OABSS change percentage is defined as dividing the difference between preoperative and postoperative OABSS by preoperative OABSS, which varies from 0 to 15. If the score is over 50%, the treatment will be considered as effective.